CLINICAL TRIAL: NCT06424080
Title: Oncological and Perioperative Outcomes of Laparoscopic Versus Robotic Partial Nephrectomy for Treatment of Renal Tumors.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Hossam Kandeel, Yassin Abdelghaffar st-from Gamal Abdel Nasar st- faculty of medicine, Menoufia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6-2024UROL12
Record Dates: First submitted 2024-05-13; First posted 2024-05-21 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic partial nephrectomy (Other): cases of renal cell carcinoma , localized tumors , candidate for laparoscopic partial nephrectomy
  Interventions: Procedure: laparoscopic partial nephrectomy
- robotic partial nephrectomy (Other): cases of renal cell carcinoma , localized tumors , candidate for robotic partial nephrectomy
  Interventions: Procedure: robotic partial nephrectomy

INTERVENTIONS:
Procedure: laparoscopic partial nephrectomy — cases amenable for partial nephrectomy
  Arms: laparoscopic partial nephrectomy
Procedure: robotic partial nephrectomy — cases amenable for partial nephrectomy
  Arms: robotic partial nephrectomy

SUMMARY:
partial nephrectomy offers lower renal function impairment and equivalent oncological survival outcomes compared with radical nephrectomy in those with T1 tumors.

As urology has embraced the gradual shift from open to minimally invasive surgery (MIS), PN is being completed more often by laparoscopic and robotic methods .

The first laparoscopic transperitoneal partial nephrectomy was reported in 1993 by Winfield, with the retroperitoneal approach introduced 1 year later With advancing robotic technology and the development of the DaVinci system, urologists began to explore the realm of robotic-assisted urologic surgery. In 2004, Gettman et al. published a paper describing their experience with robotic-assisted laparoscopic partial nephrectomy.

Moreover, robotic assisted partial nephrectomy (RAPN) and laparoscopic partial nephrectomy (LPN) seems to be significantly better than OPN in terms of perioperative complications, estimated blood loss and hospital stay. Conversely, transfusion rate, ischemia time, change in estimated glomerular filtration rate and early cancer outcomes are similar between the two approaches. International guidelines recommend the use of both approaches according to the surgeon and patient preferences.

so, we are plaining to do the study comparing between RAPN and LPN regarding feasibility and ability of both techniques.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) represents a significant burden of malignancy. Over the past 2-3 decades, the incidence of kidney cancer has steadily increased all around the world ,.The EUA Guidelines suggested that surgery is the only curative treatment for localized renal cell carcinoma.

Surgical treatment of RCC either radical or partial nephrectomy is related to the clinical stage of the disease and to the general condition of the patient. Modern medical imaging has further revolutionized the role of PN due to the increasing volume of incidentally diagnosed small renal masses.

Indeed, partial nephrectomy offers lower renal function impairment and equivalent oncological survival outcomes compared with radical nephrectomy in those with T1 tumors.

As urology has embraced the gradual shift from open to minimally invasive surgery (MIS), PN is being completed more often by laparoscopic and robotic methods .

The first laparoscopic transperitoneal partial nephrectomy was reported in 1993 by Winfield, with the retroperitoneal approach introduced 1 year later With advancing robotic technology and the development of the DaVinci system, urologists began to explore the realm of robotic-assisted urologic surgery. In 2004, Gettman et al. published a paper describing their experience with robotic-assisted laparoscopic partial nephrectomy.

Moreover, robotic assisted partial nephrectomy (RAPN) and laparoscopic partial nephrectomy (LPN) seems to be significantly better than OPN in terms of perioperative complications, estimated blood loss and hospital stay. Conversely, transfusion rate, ischemia time, change in estimated glomerular filtration rate and early cancer outcomes are similar between the two approaches. International guidelines recommend the use of both approaches according to the surgeon and patient preferences.

so, we are plaining to do the study comparing between RAPN and LPN regarding feasibility and ability of both techniques.

ELIGIBILITY:
Inclusion Criteria:

* renal mass T1 according to TNM amenable for partial nephrectomy.

Exclusion Criteria:

* any unfit pt for partial nephrectomy
* more than 7cm tumor
* mass not amenable for partial nephrectomy
* metastatic tumor or locally advanced

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
to compare between laparoscopic and robotic partial nephrectomy regards ischemia time | 1 year
  to compare between laparoscopic and robotic partial nephrectomy regards ischemia time

SECONDARY OUTCOMES:
compare between laparoscopic and robotic partial nephrectomy pathological safty margin | 1 year
  compare between laparoscopic and robotic partial nephrectomy pathological safty margin

CONTACTS AND LOCATIONS:
Overall Officials: hossam elsayed kandeel, MSC, Study Director — Director
Locations (1):
- Hossam Kandeel, Shibīn al Kawm, Menoufia -, Egypt